CLINICAL TRIAL: NCT01170845
Title: A Pilot Study of Effect of Neutrophil Elastase Inhibitor on Lung Injury After Esophagectomy
Brief Title: Effect of Neutrophil Elastase Inhibitor on Lung Injury After Esophagectomy
Acronym: NEIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Institutional Review Board, Yokohama City University, Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 531
Record Dates: First submitted 2010-07-23; First posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2007-03

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; Postoperative respiratory complications; neutrophil elastase inhibitor
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): Patients in the control group received saline for 7 days starting at the beginning of surgery
  Interventions: Drug: sivelestat sodium hydrate
- S group (Active Comparator): Patients in the S group received sivelestat sodium hydrate at a dosage 4.8mg/kg/day for 7 days starting at the beginning of surgery
  Interventions: Drug: sivelestat sodium hydrate

INTERVENTIONS:
Drug: sivelestat sodium hydrate — saline or sivelestat sodium hydrate intravenously for 7 days starting the beginning of surgery
  Other Names: Elaspol

SUMMARY:
A neutrophil elastase inhibitor may have effect on suppression of the lung injury after thoransthoracic esophagectomy. The investigators hypothesized that postoperative complication, particularly respiratory complication may be reduced by neutrophil elastase inhibitor after esophagectomy.

DETAILED DESCRIPTION:
The aim of this study was to clarify the usefulness of perioperative administration of sivelestat sodium hydrate, a selective inhibitor of neutrophil elastase in the pulmonary function, systemic inflammatory response, and the postoperative clinical course following video-assisted thoracoscopic esohpagectomy for esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic esophageal squamous cell carcinoma

Exclusion Criteria:

* Preoperative chemoradiotherapy
* Cardiovascular disease with NYHA grade III or IV
* Pulmonary disorder with Hugh-Jones classification II, III, IV, or V, preo
* Liver cirrhosis
* Renal failure

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 9 days
  the arterial oxygen pressure

SECONDARY OUTCOMES:
Pulmonary function | 9 days
  fraction of inspired oxygen ratio (PF ratio)
Pulmonary function | 9 days
  the duration of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Chikara Kunisaki, MD,PhD, Study Chair — Yokohama City University Medical Center
Locations (1):
- Chikara Kunisaki, Yokohama, Kanagawa, Japan

REFERENCES:
- [Derived] Makino H, Kunisaki C, Kosaka T, Akiyama H, Morita S, Endo I. Perioperative use of a neutrophil elastase inhibitor in video-assisted thoracoscopic oesophagectomy for cancer. Br J Surg. 2011 Jul;98(7):975-82. doi: 10.1002/bjs.7499. Epub 2011 May 9. PMID 21557207